CLINICAL TRIAL: NCT07302906
Title: The SOAR Trial (Scribe Optimization for Ambulatory Records): Ambient Artificial Intelligence Scribe With Voa Health for Generating Medical Documentation From Outpatient Visit Audio - A Randomized Controlled Trial
Brief Title: Randomized Trial of an Ambient AI Scribe (Voa Health) That Converts Outpatient Visit Audio Into Draft Notes, Comparing Visits With vs. Without AI Across Multiple Clinics to Assess Physician Well-being, Documentation Burden and Patient Experience.
Acronym: SOAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Angelo Basei de Paula (Other)
Collaborators: Universidade Federal do Paraná (Other)
Responsible Party: Sponsor-Investigator, Pedro Angelo Basei de Paula, Research Coordinator, Universidade Federal do Paraná
Organization: Universidade Federal do Paraná (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SOAR-UFPR-VOA-001; 81736024.4.0000.0096 (Other Grant/Funding Number: Research Ethics Committee for Human Subjects - Health Sciences Sector, Federal University of Paraná (UFPR)); 51.562.244/0001-07 (Other Grant/Funding Number: Voa Health)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Burnout, Professionals; Medical Records Systems, Computerized; Physician-Patient Relations; Ambulatory Care
Keywords: ambient AI scribe; artificial intelligence; clinical documentation; medical note generation; electronic health record; physician well-being; documentation burden; patient experience; outpatient clinics; randomized controlled trial
MeSH Terms: conditions — Burnout, Psychological | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment at the level of individual consultations. Each eligible visit is randomized to either usual documentation (without AI) or documentation assisted by the ambient AI scribe. Each patient contributes only one study consultation to a single arm.
Masking Description: Open-label pragmatic trial; physicians and patients are aware of the use of the AI scribe
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient AI scribe (Voa Health) (Experimental): Outpatient consultations in which the Voa Health ambient AI scribe is active. The system records the audio of the visit and generates a structured draft clinical note based on specialty-specific templates. The physician reviews, edits, and signs the note in the EMR. After the visit, the physician and the patient complete brief questionnaires about workload, well-being, communication, empathy, and satisfaction.
  Interventions: Other: Ambient AI scribe for clinical documentation (Voa Health)
- Usual documentation without AI scribe (Active Comparator): Outpatient consultations in which documentation is performed using usual methods without AI support (standard clinical practice). Audio of the visit may be recorded for study purposes, but no AI-generated note is shown to the clinician. After the visit, the physician and the patient complete the same brief questionnaires about workload, well-being, communication, empathy, and satisfaction.
  Interventions: Other: Usual documentation without AI scribe (standard care)

INTERVENTIONS:
Other: Ambient AI scribe for clinical documentation (Voa Health) — Use of an ambient artificial-intelligence (AI) scribe during outpatient consultations. The Voa Health system records the audio of the visit and generates a structured draft clinical note based on specialty-specific templates that follow the usual flow of each clinic. After the consultation, the physician reviews, edits, and signs the note in the electronic medical record. The AI does not make diagnostic or therapeutic decisions; it only assists documentation. All other aspects of clinical care follow routine practice.
  Arms: Ambient AI scribe (Voa Health)
Other: Usual documentation without AI scribe (standard care) — Clinical documentation performed using usual methods without AI support (standard care). Physicians document the encounter in the electronic medical record as they normally do (typing, dictation, or handwritten notes as applicable). Audio of the visit may be recorded for study purposes, but no AI-generated draft note is shown to the clinician. After the consultation, physicians and patients complete the same brief questionnaires about workload, well-being, communication, empathy, and satisfaction.
  Arms: Usual documentation without AI scribe

SUMMARY:
The goal of this randomized clinical trial is to learn whether an "ambient AI scribe" (Voa Health) can reduce documentation burden and improve physician well-being and patient experience in outpatient clinics. The AI scribe listens to the audio of the consultation and produces a draft of the clinical note that the physician reviews and edits.

In this study, consultations are randomized to 2 groups: usual documentation (without AI) or documentation assisted by the AI scribe. Adult patients seen in participating clinics, and their physicians, are invited to take part. For both groups, the consultation audio is recorded and, at the end of the visit, physicians and patients complete short questionnaires about well-being, workload, communication, empathy, and satisfaction. The questionnaires are based on internationally used scales (such as PFI, Mini-Z, NASA-TLX, CARE, PSQ-18, and CAT) but adapted to keep them brief and feasible in routine care.

The main questions are whether the AI scribe lowers the time and effort needed to document the visit, improves physician professional fulfillment and reduces burnout, and whether it affects how patients perceive the communication, empathy, and overall quality of the consultation. No drugs or devices are being tested. The results are expected to guide hospitals on the safe and effective use of ambient AI scribes in real-world clinical practice.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to assess the impact of an ambient artificial-intelligence (AI) scribe on physician well-being, documentation workload, and patient experience in routine outpatient care.

The intervention consists of using the Voa Health ambient AI scribe during clinical encounters. The system records the audio of the consultation and generates a structured draft clinical note in real time, aligned with specialty-specific templates that reflect the routine workflow of each clinic (for example, different templates for general cardiology, heart failure, dyslipidemia, etc.). At the end of the visit, the physician reviews, edits, and signs the draft in the electronic medical record (EMR), remaining fully responsible for the accuracy and completeness of the documentation. In the control condition, physicians conduct consultations and document encounters using their usual methods without AI support. For study purposes, audio may still be recorded in the control arm, but no AI-generated note is displayed or used by the clinician.

The unit of randomization is the individual consultation. For participating physicians, eligible visits are automatically allocated to one of two parallel arms: (1) usual documentation without AI and (2) documentation assisted by the ambient AI scribe. Randomization is designed to preserve the existing organization of each clinic and to avoid interference with scheduling or patient flow. Clinical care, diagnostic and therapeutic decisions, and follow-up procedures are not dictated by the protocol and follow usual practice; the only experimental element is the use (or non-use) of the AI scribe for documentation and the collection of audio and questionnaires.

Adult patients seen in participating outpatient clinics, and their physicians, are invited to take part. After informed consent, the entire consultation is audio-recorded. Immediately after each visit, both patient and physician are asked to complete brief, structured questionnaires that capture the main outcomes of interest. To keep data collection feasible in a busy ambulatory setting, the instruments were built from subsets of items derived from internationally used scales, while keeping the number of questions per consultation small.

For physicians, items are drawn from the Professional Fulfillment Index (PFI), the Mini-Z 2.0 survey, and the 4-item Physician Task Load / NASA-TLX. These items assess professional fulfillment and burnout (physical and emotional exhaustion), perceived sufficiency of time for documentation, work in the EMR outside direct patient contact, perceived documentation burden, and temporal demand of the visit. Additional study-specific items evaluate the perceived quality and completeness of the final note, time required to edit the AI-generated draft, confidence that key clinical details were captured, occurrence of potential AI "hallucinations" (information not actually stated in the visit), and the perceived impact of documentation on attention to the patient.

For patients, questionnaires use items derived from the Consultation and Relational Empathy (CARE) Measure, the Patient Satisfaction Questionnaire Short-Form (PSQ-18), and the Communication Assessment Tool (CAT). These items cover domains such as active listening, understanding of patient concerns, clarity of explanations, adequacy of time spent with the physician, perceived empathy, overall satisfaction with care, and understanding of diagnosis and treatment. In the AI arm, one additional item specifically asks whether the use of AI during the consultation helped, did not change, or hindered the clarity of communication with the physician.

The primary outcomes are physician-reported well-being and perceived documentation workload when using the ambient AI scribe compared with usual documentation. Key secondary outcomes include patient-reported experience and satisfaction, physician-rated quality and completeness of notes, time required for documentation and for editing AI-generated drafts, and the frequency and clinical relevance of AI-related documentation errors or hallucinations. All outcomes are measured at the level of the individual consultation, immediately after each visit.

The trial is initially conducted in multiple outpatient clinics of Hospital de Clínicas of the Federal University of Paraná (UFPR), Brazil, across different medical specialties. In each service, structured note templates are developed in collaboration with local clinical leaders so that the AI-generated drafts reflect the real-world flow of that specialty without changing the standard of care. Medical students and residents trained in the protocol may support consent and questionnaire administration under supervision of attending physicians, to ensure consistent and feasible data collection.

Data are stored in secure, access-controlled servers, with linkage between audio recordings, questionnaires, and EMR notes managed through coded identifiers. A data monitoring committee, independent from the development team of the AI scribe, periodically reviews aggregated data for protocol adherence, data quality, and any safety concerns related to the use of AI in documentation (for example, systematic documentation errors that could potentially affect patient care). Because the intervention is limited to documentation support and clinicians remain responsible for all clinical decisions and for finalizing the notes, the overall risk of participation is considered minimal.

The protocol allows for future expansion to other outpatient services and collaborating centers that adopt the same randomization, data collection procedures, and outcome definitions. The results are expected to provide pragmatic evidence on how ambient AI scribes can be implemented safely and effectively in real-world clinical practice, particularly regarding their impact on physician well-being, documentation workload, and the patient's experience of the consultation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) attending participating outpatient clinics at Hospital de Clínicas - Federal University of Paraná during the study period.
* Receiving care from a physician who is participating in the trial.
* Able to understand Portuguese and provide written informed consent for audio recording of the consultation and completion of brief questionnaires.
* Able to complete the post-visit questionnaires (with assistance if needed).
* Physicians (attendings or residents) working in the participating outpatient clinics.
* Use the hospital electronic medical record in routine care.
* Agree to have their consultations audio-recorded and to complete brief post-visit questionnaires for each included visit.

Exclusion Criteria:

* Patients younger than 18 years.
* Emergency, urgent-care, or inpatient consultations.
* Patients with significant cognitive impairment, acute distress, or clinical instability that, in the opinion of the treating physician, precludes informed consent or completion of questionnaires.
* Patients under legal guardianship or otherwise unable to provide their own consent.
* Consultations in which either the patient or the physician declines audio recording or participation in the study.
* Consultations in which the AI system is unavailable or malfunctioning (for protocol adherence analyses only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Physician documentation workload during the visit | Immediately after each outpatient consultation (same day)
  Documentation workload reported by physicians immediately after the consultation, measured with an adapted 4-item Physician Task Load / NASA-TLX scale. Each item is rated on a 5-point Likert scale (very low, low, moderate, high, very high) for temporal demand, mental effort, effort required for documentation, and frustration related to documentation. A summary score (mean of item scores; higher values = greater workload) will be compared between consultations with the ambient AI scribe and consultations with usual documentation without AI.
Physician well-being / exhaustion during the visit | Immediately after each outpatient consultation (same day)
  Physician well-being during the consultation, assessed with two items derived from the Professional Fulfillment Index (PFI) for physical and emotional exhaustion. Each item is rated on a 5-point scale from 0 (not at all) to 4 (extremely). A composite exhaustion score (mean of the two items; higher values = greater exhaustion) will be compared between consultations with the ambient AI scribe and consultations with usual documentation without AI.

SECONDARY OUTCOMES:
Patient experience of communication and empathy | Immediately after each outpatient consultation (same day)
  Patient-reported experience of the consultation, including active listening, understanding of concerns, clarity of explanations, perceived empathy, time spent with the physician, and overall satisfaction. Items are derived from the CARE Measure, PSQ-18, and Communication Assessment Tool (CAT), rated on 5-point Likert scales. A composite score (mean of item scores; higher values = better experience) will be compared between consultations with the ambient AI scribe and consultations with usual documentation without AI.
Patient understanding of diagnosis and treatment | Immediately after each outpatient consultation (same day)
  Single item asking patients how much they understood about their diagnosis and treatment after the consultation, rated on a 5-point scale from 1 (nothing) to 5 (completely). Scores will be compared between consultations with the ambient AI scribe and consultations with usual documentation without AI.
Physician-rated quality and completeness of clinical notes | Immediately after finalizing documentation for each consultation (same day)
  Physician global rating of the final clinical note for the consultation (clarity, organization, and completeness), using a 5-point scale adapted from Mini-Z (poor, marginal, satisfactory, good, excellent). Scores will be compared between consultations with the ambient AI scribe and consultations with usual documentation without AI.
Time required for documentation outside direct patient contact | Immediately after each outpatient consultation (same day)
  Physician self-reported time spent working on the electronic medical record outside direct patient contact for that consultation (for example, after the patient leaves the room), including review and editing of AI-generated notes when applicable. Time is rated in ordered categories (almost none; minor edits; moderate edits; extensive edits). Distributions of categories will be compared between the ambient AI scribe and usual documentation conditions.
Proportion of consultations with AI-related hallucinations in documentation | Immediately after each AI-assisted consultation (same day)
  Among consultations in the ambient AI scribe arm, physicians indicate whether the AI inserted any information in the draft note that was not actually mentioned in the consultation. The outcome is the proportion of AI-assisted consultations with at least one reported hallucination.
Proportion of clinical notes with documentation errors in blinded external review | Within 30 days after finalizing each clinical note
  De-identified clinical notes from both study arms (AI scribe and usual documentation) will be randomly mixed and independently reviewed by at least two clinicians who are blinded to group allocation. Reviewers will classify whether each note contains any clinically relevant documentation error, including fabricated or incorrect information ("hallucinations") that does not match the plausible content of a standard outpatient visit. The primary variable is the proportion of notes with at least one such error in each arm; proportions will be compared between AI-scribe and usual documentation conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Lenci Marques, MD, PhD, Principal Investigator — Universidade Federal do Paraná; Pedro Angelo Basei de Paula, Medical Student, Study Director — Universidade Federal do Paraná

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the main published results may be shared with other researchers upon reasonable request to the principal investigator and after approval by the Hospital de Clínicas/UFPR data governance. The study protocol and statistical analysis plan will be made available as supplementary material. The analytic code (e.g., R/Python scripts) used for data cleaning and analysis will be deposited in a public Git repository (such as GitHub) after publication of the primary results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available after publication of the primary results and for at least 5 years thereafter.
Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal, subject to data-use agreement and approval by the local ethics committee/IRB and the sponsor institution. Requests should be sent to the principal investigator (Gustavo Lenci Marques, Universidade Federal do Paraná).

REFERENCES:
- [Background] Majid Afshar, M.D., M.S., Mary Ryan Baumann, Ph.D., Felice Resnik, Ph.D., Josie Hintzke, M.S., and Others. A Pragmatic Randomized Controlled Trial of Ambient Artificial Intelligence to Improve Health Practitioner Well-Being. NEJM AI. November 26, 2025;2(12)
- [Background] Grace Hong, B.A., Lauren Wilcox, Ph.D., Amelia Sattler, M.D., Samuel Thomas, M.D., Nina Gonzalez, M.D., Marissa Smith, Ph.D., John Hernandez, Ph.D., Margaret Smith, M.B.A., Steven Lin, M.D., and Robert Harrington, M.D. Clinicians' Experiences with EHR Documentation and Attitudes Toward AI-Assisted Documentation. Stanford University School of Medicine and Google Health. 2020.
- [Background] Davenport T, Kalakota R. The potential for artificial intelligence in healthcare. Future Healthc J. 2019 Jun;6(2):94-98. doi: 10.7861/futurehosp.6-2-94. PMID 31363513
- [Background] Quiroz JC, Laranjo L, Kocaballi AB, Berkovsky S, Rezazadegan D, Coiera E. Challenges of developing a digital scribe to reduce clinical documentation burden. NPJ Digit Med. 2019 Nov 22;2:114. doi: 10.1038/s41746-019-0190-1. eCollection 2019. PMID 31799422
- [Background] Cheng CG, Wu DC, Lu JC, Yu CP, Lin HL, Wang MC, Cheng CA. Restricted use of copy and paste in electronic health records potentially improves healthcare quality. Medicine (Baltimore). 2022 Jan 28;101(4):e28644. doi: 10.1097/MD.0000000000028644. PMID 35089204
- [Background] Olson KD, Meeker D, Troup M, Barker TD, Nguyen VH, Manders JB, Stults CD, Jones VG, Shah SD, Shah T, Schwamm LH. Use of Ambient AI Scribes to Reduce Administrative Burden and Professional Burnout. JAMA Netw Open. 2025 Oct 1;8(10):e2534976. doi: 10.1001/jamanetworkopen.2025.34976. PMID 41037268
- [Background] Yixing Jiang, Kameron C. Black, D.O., M.P.H., Gloria Geng, Danny Park, James Zou, Ph.D., Andrew Y. Ng, Ph.D., and Jonathan H. Chen, M.D., Ph.D. MedAgentBench: A Virtual EHR Environment to Benchmark Medical LLM Agents. NEJM AI. August 14, 2025;2(9)
- [Background] Afshar M, Resnik F, Baumann MR, Hintzke J, Lemmon K, Sullivan AG, Shah T, Stordalen A, Oberst M, Dambach J, Mrotek LA, Quinn M, Abramson K, Kleinschmidt P, Brazelton T, Twedt H, Kunstman D, Wills G, Long J, Patterson BW, Liao FJ, Rasmussen S, Burnside E, Goswami C, Gordon JE. A Novel Playbook for Pragmatic Trial Operations to Monitor and Evaluate Ambient Artificial Intelligence in Clinical Practice. NEJM AI. 2025 Sep;2(9):10.1056/aidbp2401267. doi: 10.1056/aidbp2401267. Epub 2025 Aug 28. PMID 40959192
- [Background] BASEI DE PAULA, P., BRUNETI SEVERINO, J., BERGER, M., VEIGA, M., PARENTE RIBEIRO, K., LOURES, F., TODESCHINI, S., ROEDER, E., MARQUES, G.. Improving documentation quality and patient interaction with AI: a tool for transforming medical records-an experience report. Journal of Medical Artificial Intelligence, North America, 8, jan. 2025. Available at: <https://jmai.amegroups.org/article/view/9651>
- [Background] Paul J. Lukac, M.D., M.B.A., M.S., and Others. Ambient AI Scribes in Clinical Practice: A Randomized Trial. NEJM AI. November 26, 2025;2(12)
- [Background] Eileen Kim, M.D., Vincent X. Liu, M.D., M.Sc., and Karandeep Singh, M.D., M.M.Sc. AI Scribes Are Not Productivity Tools (Yet). NEJM AI. November 26, 2025;2(12)